CLINICAL TRIAL: NCT03009656
Title: Assessing Accuracy of Clinical Diagnosis and Lesion Location in Acute Neurological Deficits - How Good Are Neurologists?
Acronym: HOGAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-01819
Record Dates: First submitted 2017-01-02; First posted 2017-01-04 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Stroke Syndrome; Stroke Hemorrhagic; Stroke, Acute; Strokes Thrombotic; Emergencies; Diagnostic Self Evaluation
Keywords: Stroke; Emergency; Focal Neurological Deficits; Diagnostic
MeSH Terms: conditions — Stroke; Hemorrhagic Stroke; Thrombotic Stroke; Emergencies; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No study specific interventions

SUMMARY:
The emergency setting for acute neurological conditions, such as stroke, is peculiar due to time pressure and limited resources for further diagnostics. Clinical skills are essential for swift and accurate bedside diagnosis and thus are the basis for early and correct treatment. This is especially evident in the context of computed tomography being the standard neuroimaging method world-wide with its limitations for detecting smaller infarcts, strokes in the posterior fossa and reduced sensitivity for stroke mimics, such as epileptic seizures or migraine aura. To date, the accuracy of clinical bedside diagnosis of stroke by neurologists verified by magnetic resonance imaging (MRI) in the emergency setting has not been studied in detail. In order to improve clinical diagnosing and future treatment it is essential to quantify the accuracy of clinical diagnosis of stroke in the emergency setting ("how good are neurologists?") and to assesses whether there are any differences between experienced staff neurologists and junior physicians.

DETAILED DESCRIPTION:
Background:

The emergency setting for acute neurological conditions, such as stroke, is peculiar due to time pressure and limited resources for further diagnostics. Clinical skills are essential for swift and accurate bedside diagnosis and thus are the basis for early and correct treatment. This is especially evident in the context of computed tomography being the standard neuroimaging method world-wide with its limitations for detecting smaller infarcts, strokes in the posterior fossa and reduced sensitivity for stroke mimics, such as epileptic seizures or migraine aura. To date, the accuracy of clinical bedside diagnosis of stroke by neurologists verified by magnetic resonance imaging (MRI) in the emergency setting has not been studied in detail. Management of acute stroke patients is a main interest of the neurovascular research group at Inselspital Bern. For example, the investigators analysed the prediction of large vessel occlusion in acute stroke patients by clinical examination and found a significant association of stroke severity measured with the NIHSS score and location of vessel occlusion. Analysis of outcome in stroke patients with mild and rapidly improving symptoms demonstrated that three of four of these patients had a favourable outcome, but those with a central vessel occlusion were likely to deteriorate with poor outcome. These studies showed that there is a correlation of clinical symptoms with the mechanism of stroke, which is important for the outcome after treatment. Importantly, however, the quality of clinical assessment itself is likely highly variable, for example depending on the experience of the treating physician. Factors influencing this clinical assessment, which needs to be done under high temporal and emotional pressure in the emergency setting have not been investigated so far but might be crucial for rapid and successful treatment ("time is brain").In order to improve clinical diagnosing and future treatment it is essential to quantify the accuracy of clinical diagnosis of stroke in the emergency setting ("how good are neurologists?") and to assesses whether there are any differences between experienced staff neurologists and junior physicians.

Rationale:

By assessing whether prediction of aetiology of acute neurological deficits is experience-based the investigators aim to understand what symptoms/signs impede the in-experienced from swiftly making the correct diagnosis in the emergency setting. This should help to improve resident training and with this treatment of patients with acute neurological deficits.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Non-refusal of "general consent"
* Patients with focal clinical neurological deficits with symptom onset of < 6 hours or wake-up strokes.

Exclusion Criteria:

* Interval from symptom onset to clinical examination of > 6 hours.
* Patients who do not have focal clinical neurological deficit at examination will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with focal neurological deficits in the Emergency Room of Inselspital Bern.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2017-01-10 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of correct initial diagnoses by emergency physicians in patients with focal clinical neurological deficits | 7 days +/- 7 days
  Primary endpoint is the proportion of correct initial diagnoses by emergency physicians in patients with focal clinical neurological deficits, calculated by comparing the initial assessment with the final diagnosis at discharge. If the initial assessment was correct, the diagnosis of the emergency physician will be rated as correct (correct answer = Ac), if it was incorrect, it will be rated as incorrect (incorrect answer = Ai).
  The proportion of accurate initial diagnoses will be calculated as:
  Ac / (Ac + Ai)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Schankin, PD Dr. med., Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Bern University Hospital - Inselspital, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No